CLINICAL TRIAL: NCT04286906
Title: Multidimensional Assessment of Dyspnea in Asthma
Acronym: MIDAS
Status: Terminated | Type: Observational
Why Stopped: greatly reduced active file of potentially includible patients
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_11; 2019-A02795-52 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-02-21; First posted 2020-02-27 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Asthma
Keywords: Asthma; Breathlessness
MeSH Terms: conditions — Asthma; Dyspnea | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One group (cohort): Asthmatic patients
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — MultiDimensional Profile (MDP), Anxiety-Depression Hospital Scale (HADs), Nijmegen

SUMMARY:
Breathlessness is a symptom of asthma that occurs in relation with lower airway obstruction. However, this sensation is not specific of asthma and may be the expression of other disorders. In particular, it can testify to anxiety or hyperventilation, two disorders frequently associated with asthma. The systematic interpretation of dyspnea as a manifestation of asthma in asthmatic patients may lead to an inappropriate increase in asthma controllers.

Identifying the cause of dyspnea in asthmatic patients (airway obstruction, anxiety or hyperventilation) is therefore crucial for the clinician.

This could be facilitated by a multidimensional assessment of dyspnea, evaluating the kind of sensation felt by the patient (for example chest tightness, air hunger etc.) and emotions associated to respiratory sensations (for example anxiety, fear etc.).

The objectives of this project are to assess: (1) the sensory and affective dimensions of dyspnea in asthma and, (2) their connection to asthma control, anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of asthma confirmed by:

   * A history of symptoms compatible with asthma
   * AND a history of airway obstruction, according to the GINA definition (2017): FEV1/FVC ratio lower than the lower limit of the predicted value at baseline or after a bronchial provocation test
   * AND a variability of airway obstruction defined by at least one of the following criteria:

   oReversibility of airway obstruction after bronchodilators (400 µg of salbutamol): FEV 1 increases by> 200 mL and> 12% compared to baseline
   * OR delta peak-flow over the day / average peak-flow averaged over 2 weeks> 10%
   * OR variability in FEV1 between two visits> 200 mL and> 12%
   * OR an increase in FEV1 of> 200 mL and> 12% compared to the baseline after 4 weeks of treatment with oral corticosteroids
   * OR a positive methacholine challenge: decrease in FEV1 by more than 20% for a dose <1600 µg
2. Experience of dyspnea in the past 7 days
3. Age> 18 years old
4. Social protection affiliation 5. Written informed consent

Exclusion Criteria:

1. Age <18 years old
2. Active smoker or quitting smoking for less than a year
3. Severe exacerbation or respiratory infection within 4 weeks before inclusion (severe exacerbation is defined by an increase in systemic corticosteroid therapy for at least 3 days or injection of a single dose of delayed corticosteroid, emergency room visit due to asthma (with systemic corticosteroid therapy), or hospitalization due to asthma).
4. Inability to respond to questionnaires for any reason
5. Presence of any pathology other than asthma which may be responsible for dyspnea, in particular cardiovascular or respiratory (ischemic heart disease, heart failure, chronic obstructive pulmonary disease, diffuse interstitial pneumonitis, lung cancer, non-exhaustive list) with the exception of anxiety and hyperventilation syndrome
6. Pregnancy
7. Persons under guardianship
8. Refusal to sign consent or participate in the study
9. No social protection affiliation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Asthmatic patients reporting breathlessness
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Description of the sensory and affective dimensions of dyspnea | At baseline
  MultiDimensional Profile (MDP) scores QS and A2

SECONDARY OUTCOMES:
Association between dyspnea intensity and asthma control | At baseline
  Correlation between MDP scores QS and A2 and ACQ-5 Correlation between MDP scores QS and A2 and ACQ-5
Association between dyspnea intensity and anxiety | At baseline
  Correlation between MDP scores QS and A2 and anxiety score HAD-A
Association between dyspnea intensity and hyperventilation | At baseline
  Correlation between MDP scores QS and A2 and the Nijmegen score
Association between change in dyspnea intensity and in asthma control | Difference between baseline and 6 months
  Correlation between change in MDP scores QS and A2 and change in ACQ-5
Association between change in dyspnea intensity and in anxiety | Difference between baseline and 6 months
  Correlation between change in MDP scores QS and A2 and change in HAD-A score
Association between change in dyspnea intensity and in hyperventilation | Difference between baseline and 6 months
  Correlation between change in MDP scores QS and A2 and change in the Nijmegen score

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Chenivesse, MD PhD, Principal Investigator — CHU Lille
Locations (5):
- France (5):
  - Ch Dunkerque, Dunkirk
  - Hopital Saint Vincent - Saint Antoine - Lille, Lille
  - Hop Calmette Chu Lille, Lille
  - Hu Paris Nord Site Bichat Aphp - Paris 18, Paris
  - Hu Paris Sud Site Kremlin Bicetre Aphp - Le Kremlin Bicetre, Paris

IPD SHARING:
Plan to Share IPD: No